CLINICAL TRIAL: NCT03016936
Title: MET: REevaluation for Perioperative cArdIac Risk (MET-REPAIR) Observational Multicentre Study
Brief Title: MET: REevaluation for Perioperative cArdIac Risk (MET-REPAIR)
Acronym: MET-REPAIR
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: MET-REPAIR
Record Dates: First submitted 2016-10-26; First posted 2017-01-11 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Non Cardiac Surgery
Keywords: Metabolic equivalents (METs); European Society of Anaesthesiology (ESA); Noncardiac surgery; Cardiovascular Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the NTproBNP sub-study, 5 ml of blood is sampled. No storage after measurement.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subgroup for NTproBNP Substudy: Planned subgroup analyses in patients undergoing vascular, orthopaedic, thoracic surgery, and in patients aged 65 years or older with a RCRI <2 and NSQIP- MICA <1%

SUMMARY:
Multicentre international prospective cohort study designed to answer the question: "In patients undergoing elevated risk noncardiac surgery, are METs estimated by questionnaire associated with perioperative major adverse cardiovascular events or cardiovascular mortality?" If so:

1. What is the optimal cut-off for METs estimated by questionnaire to predict perioperative major adverse cardiovascular events or cardiovascular mortality?
2. How does the optimal cut-off compare with the currently guideline-endorsed 4-MET cut-off?

DETAILED DESCRIPTION:
In spite of scarce and non-conclusive evidence on the prognostic value of self-reported functional capacity for perioperative cardiovascular events, the estimation of cardiovascular functional capacity in metabolic equivalents (METs) based on a questionnaire represent the core question in the preoperative cardiac risk assessment in patients undergoing elevated risk noncardiac surgery endorsed by ESA, the ESC, and the ACC/AHA. MET-REPAIR will examine the ability of MET estimated using a questionnaire to predict perioperative cardiovascular events correcting for preoperative risk factors, (e.g. comorbidity and type of surgery) and calculate the effect on risk stratification (net reclassification improvement) by the addition of METs estimated by questionnaire to established risk scores, such as the Revised Cardiac Risk Score (Lee-index) and the NSQIP MICA . Further, investigators will address alternative approaches to functional capacity estimation (1. ability to climb stairs; 2. self-assessed functional capacity compared to peers; 3. Daily/weekly physical activity) and their predictive value for perioperative cardiovascular events.

The association between elevated natriuretic peptides prior to noncardiac surgery and perioperative cardiovascular events is well established. However, a direct comparison of the predictive ability of biomarkers vs. self-reported MET is lacking. Therefore, in a substudy (NTproBNP substudy), investigators will evaluate in how far the addition of NTproBNP improve prediction of perioperative cardiovascular events and cardiovascular mortality when added to clinical data and estimated METs.

ELIGIBILITY:
Inclusion Criteria:

* Planned as Inpatients after surgery
* 45 years of age or older AND undergoing elective elevated-risk noncardiac surgery as defined by either a Revised Cardiac Risk Index ≥ 2 [9] OR NSQIP MICA>1% [10]
* 65 years of age or older and undergoing intermediate or high-risk procedures [3]
* Signed Written informed consent

Exclusion Criteria:

* Non-elective surgery, i.e. planned to occur ≤ 72 hours after diagnosis of the acute condition that makes the procedure necessary
* Acute coronary syndrome or uncontrolled congestive heart failure within the last 30 days of planned day of surgery
* Stroke within the last 7 days of planned day of surgery
* Outpatients
* Patients unable to perform ambulation due to congenital or longstanding illnesses/states (e.g. paraplegics, polio, etc; but explicitly not patients with fractures, needing hip replacement, etc.)
* Unable to consent or unwilling to participate
* Previous enrolment in MET REPAIR (in case of repeated surgery)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective, elevated-risk noncardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Composite of intra or postoperative inhospital cardiovascular mortality, nonfatal cardiac arrest, acute myocardial infarction, stroke and congestive heart failure requiring transfer to a higher care unit or prolonging stay on ICU/intermediate care (≥24h) | within 24 hours after surgery
  Composite of intra- or postoperative inhospital cardiovascular mortality, nonfatal cardiac arrest, acute myocardial infarction, stroke, and congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care (≥24h).

SECONDARY OUTCOMES:
composite of intra- or postoperative inhospital cardiovascular mortality, nonfatal cardiac arrest, acute myocardial infarction, stroke, and congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/IMC (≥24h) | at 30days after surgery or on discharge
  composite of intra- or postoperative inhospital cardiovascular mortality, nonfatal cardiac arrest, acute myocardial infarction, stroke, and congestive heart failure requiring transfer to a higher unit of care or prolonging stay on ICU/intermediate care (≥24h)
Inhospital all-cause mortality | at 30days after surgery
complications ≥ 3 in Clavien Dindo Classification | From date of surgery until up to day 30 after surgery or until discharge if occurred before day 30 and no follow-up call is carried out.
length of In hospital stay (days), length of ICU stay (days in the ICU) | from date of surgery until discharge or until day 30 after surgery, whichever occurs first. .
myocardial injury after noncardiac surgery (MINS) | From date of surgery until up to day 30 after surgery or until discharge if occurred before day 30 and no follow-up call is carried out.
  Only applicable for patients from centres routinely implementing a perioperative troponin screening

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Lurati Buse, PD Dr., Study Chair — Heinrich-Heine University, Duesseldorf
Locations (1):
- Universitätsklinikum Düsseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Devereaux PJ, Mrkobrada M, Sessler DI, Leslie K, Alonso-Coello P, Kurz A, Villar JC, Sigamani A, Biccard BM, Meyhoff CS, Parlow JL, Guyatt G, Robinson A, Garg AX, Rodseth RN, Botto F, Lurati Buse G, Xavier D, Chan MT, Tiboni M, Cook D, Kumar PA, Forget P, Malaga G, Fleischmann E, Amir M, Eikelboom J, Mizera R, Torres D, Wang CY, VanHelder T, Paniagua P, Berwanger O, Srinathan S, Graham M, Pasin L, Le Manach Y, Gao P, Pogue J, Whitlock R, Lamy A, Kearon C, Baigent C, Chow C, Pettit S, Chrolavicius S, Yusuf S; POISE-2 Investigators. Aspirin in patients undergoing noncardiac surgery. N Engl J Med. 2014 Apr 17;370(16):1494-503. doi: 10.1056/NEJMoa1401105. Epub 2014 Mar 31. PMID 24679062
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, De Hert S, Ford I, Gonzalez Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luescher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Uva MS, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur J Anaesthesiol. 2014 Oct;31(10):517-73. doi: 10.1097/EJA.0000000000000150. No abstract available. PMID 25127426
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, Hert SD, Ford I, Gonzalez-Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luscher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Sousa-Uva M, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur Heart J. 2014 Sep 14;35(35):2383-431. doi: 10.1093/eurheartj/ehu282. Epub 2014 Aug 1. No abstract available. PMID 25086026
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN; American College of Cardiology; American Heart Association. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines. J Am Coll Cardiol. 2014 Dec 9;64(22):e77-137. doi: 10.1016/j.jacc.2014.07.944. Epub 2014 Aug 1. No abstract available. PMID 25091544
- [Background] Holtermann A, Marott JL, Gyntelberg F, Sogaard K, Mortensen OS, Prescott E, Schnohr P. Self-reported cardiorespiratory fitness: prediction and classification of risk of cardiovascular disease mortality and longevity--a prospective investigation in the Copenhagen City Heart Study. J Am Heart Assoc. 2015 Jan 27;4(1):e001495. doi: 10.1161/JAHA.114.001495. PMID 25628408
- [Background] Stamatakis E, Hamer M, O'Donovan G, Batty GD, Kivimaki M. A non-exercise testing method for estimating cardiorespiratory fitness: associations with all-cause and cardiovascular mortality in a pooled analysis of eight population-based cohorts. Eur Heart J. 2013 Mar;34(10):750-8. doi: 10.1093/eurheartj/ehs097. Epub 2012 May 3. PMID 22555215
- [Background] Lee TH, Marcantonio ER, Mangione CM, Thomas EJ, Polanczyk CA, Cook EF, Sugarbaker DJ, Donaldson MC, Poss R, Ho KK, Ludwig LE, Pedan A, Goldman L. Derivation and prospective validation of a simple index for prediction of cardiac risk of major noncardiac surgery. Circulation. 1999 Sep 7;100(10):1043-9. doi: 10.1161/01.cir.100.10.1043. PMID 10477528
- [Background] Gupta PK, Gupta H, Sundaram A, Kaushik M, Fang X, Miller WJ, Esterbrooks DJ, Hunter CB, Pipinos II, Johanning JM, Lynch TG, Forse RA, Mohiuddin SM, Mooss AN. Development and validation of a risk calculator for prediction of cardiac risk after surgery. Circulation. 2011 Jul 26;124(4):381-7. doi: 10.1161/CIRCULATIONAHA.110.015701. Epub 2011 Jul 5. PMID 21730309
- [Derived] Stroda A, Sulot T, Roth S, M'Pembele R, Mauermann E, Ionescu D, Szczeklik W, De Hert S, Filipovic M, Beck Schimmer B, Spadaro S, Matute P, Turhan SC, van Waes J, Lagarto F, Theodoraki K, Gupta A, Gillmann HJ, Guzzetti L, Kotfis K, Larmann J, Corneci D, Howell SJ, Lurati Buse G; and the MET-REPAIR investigators. Factors affecting adherence to recommendations on pre-operative cardiac testing: A cohort study. Eur J Anaesthesiol. 2024 Sep 1;41(9):695-704. doi: 10.1097/EJA.0000000000002039. Epub 2024 Jul 10. PMID 38988248
- [Derived] Lurati Buse G, Larmann J, Gillmann HJ, Kotfis K, Ganter MT, Bolliger D, Filipovic M, Guzzetti L, Chammartin F, Mauermann E, Ionescu D, Szczeklik W, De Hert S, Beck-Schimmer B, Howell SJ; METREPAIR NTproBNP Subcohort Investigators. NT-proBNP or Self-Reported Functional Capacity in Estimating Risk of Cardiovascular Events After Noncardiac Surgery. JAMA Netw Open. 2023 Nov 1;6(11):e2342527. doi: 10.1001/jamanetworkopen.2023.42527. PMID 37938844
- [Derived] Lurati Buse GA, Mauermann E, Ionescu D, Szczeklik W, De Hert S, Filipovic M, Beck-Schimmer B, Spadaro S, Matute P, Bolliger D, Turhan SC, van Waes J, Lagarto F, Theodoraki K, Gupta A, Gillmann HJ, Guzzetti L, Kotfis K, Wulf H, Larmann J, Corneci D, Chammartin-Basnet F, Howell SJ; MET: Reevaluation for Perioperative Cardiac Risk investigators; European Society of Anaesthesiology and Intensive Care. Risk assessment for major adverse cardiovascular events after noncardiac surgery using self-reported functional capacity: international prospective cohort study. Br J Anaesth. 2023 Jun;130(6):655-665. doi: 10.1016/j.bja.2023.02.030. Epub 2023 Apr 1. PMID 37012173